CLINICAL TRIAL: NCT04227093
Title: Acetazolamide as add-on Therapy to Obstructive Sleep Apnea Surgery (ACTOS): a Parallel-group, Double-blind, Placebo-controlled, Randomized Trial
Brief Title: Acetazolamide Add-On Therapy to OSA Surgery
Acronym: ACTOS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Olivier Vanderveken, Professor and Chair Otorhinolaryngology, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B300201942507
Record Dates: First submitted 2019-12-20; First posted 2020-01-13 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Obstructive Sleep Apnea
Keywords: Acetazolamide; Carbonic anhydrase inhibitor; Upper airway stimulation; Surgery
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Acetazolamide

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acetazolamide (Active Comparator): Acetazolamide will be prescribed in unembellished white capsules of 250 mg. The drug will be administered twice daily in the morning and evening (approximately one hour before bedtime). The total treatment length will amount to 16 weeks. In case of side effects hampering treatment adherence, the daily dosage will be reduced to a single evening dose of 250 mg.
  Interventions: Drug: Acetazolamide
- Placebo (Placebo Comparator): The placebo regimen will be identical.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetazolamide — Oral acetazolamide tablets of 250 mg taken twice daily.
  Other Names: Diamox; ATC code: S01EC01
  Arms: Acetazolamide
Drug: Placebo — Matching placebo tablets taken twice daily.
  Arms: Placebo

SUMMARY:
Surgical procedures are routinely performed as an alternative to continuous positive airway pressure treatment in patients with obstructive sleep apnea (OSA). However, the response to surgery is often variable. Instability of the respiratory control during sleep (or high loop gain) has been associated with poor surgical results in previous research. Acetazolamide (AZM), a carbonic anhydrase inhibitor, has shown potential in reducing loop gain without affecting other physiological OSA traits. In this protocol the investigators will evaluate the clinical efficacy of AZM add-on therapy to surgical procedures in patients with OSA.

DETAILED DESCRIPTION:
Seventy-four patients with diagnosed moderate to severe OSA will be equally (1:1) randomized to AZM (250 mg twice daily) or placebo add-on therapy after surgery. Two surgical procedures will be performed throughout the study: barbed reposition pharyngoplasty (BRP) and upper airway stimulation (UAS) using electrical neurostimulation of the hypoglossal nerve.

Treatment allocation will occur after a satisfactory recovery in patients undergoing BRP and after titration of the device settings in patients treated with UAS. Treatment outcome will be assessed approximately 10 weeks thereafter by in-laboratory polysomnography. Two on-site follow-up visits will be scheduled to assess adherence and adverse events. The maximum treatment duration per participant will amount to 16 weeks.

Besides the aforementioned core clinical part, the study protocol will also include an optional exploratory part prior to surgery, assessing the physiological OSA traits and airflow features by means of polysomnography and drug-induced sleep endoscopy research measurements.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe OSA (i.e. 15≤ AHI <65 events per hour)
* Eligibility for either BRP or UAS surgery
* Fitness for general anesthesia (ASA ≤2)
* Capability of giving informed consent and willingness to undergo surgery

Exclusion Criteria:

* Craniofacial anomalies affecting the UA
* Body mass index (BMI) >35 kg/m²
* General contra-indications for surgery
* Central sleep apnea (defined as central AHI ≥5 events per hour)
* Contra-indications related to acetazolamide treatment

  * Hypersensitivity to sulfonamides or acetazolamide
  * Renal impairment (eGFR <60 ml/min/1.73m²), electrolyte imbalances (sodium levels <135 mmol/L or potassium levels <3.5 mmol/L) and/or adrenocortical insufficiency
  * Clinically significant neurological, metabolic (including diabetes mellitus type 1 or 2), hepatic (alanine transaminase or aspartate transaminase >2 times the upper limit of normal) and/or hematological disease
  * Chronic obstructive pulmonary disease
  * Closed-angle glaucoma
  * Professional driving or handling complex machinery due to the potential risk of exaggerated daytime sleepiness
* Concomitant intake of drugs that influence breathing, sleep, arousal and/or muscle physiology
* Inability of the patient to understand and/or comply to the study procedures
* Active psychiatric disease (psychotic illness, major depression, anxiety attacks, and alcohol or drug abuse) which prevents compliance with the requirements of the research setting
* Pregnancy or willing to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-04-22 (Actual); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) | 10 weeks of add-on therapy
  Change in AHI (events/h) from baseline to follow-up. The AHI is an index of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow).

SECONDARY OUTCOMES:
Oxygen desaturation index (ODI) | 10 weeks of add-on therapy
  Change in ODI (events/h) from baseline to follow-up. The ODI represents the average number of desaturation episodes (≥3%) per hour sleep.
Oxygen saturation (SaO2) | 10 weeks of add-on therapy
  Change in mean and minimal SaO2 (%) from baseline to follow-up.
Changes in daytime sleepiness measured with the Epworth Sleepiness Scale (ESS) | 16 weeks of add-on therapy
  The questionnaire asks subjects to rate their probability of falling asleep on a scale from 0 to 3 for eight different situations that most people encounter in their daily lives. The scores for the eight questions are added together to obtain a single number (0-24). An ESS score higher than 10 indicates the presence of excessive daytime sleepiness.
Changes in sleep-related quality of life measured with the Functional Outcome of Sleep Questionnaire (FOSQ-10) | 16 weeks of add-on therapy
  This questionnaire is an abbreviated version of the original 30-item version. The FOSQ-10 consists of 10 items that are distributed among 5 subscales: general productivity (2 items), activity level (3 items), vigilance (3 items), social outcomes (1 item), and intimacy and sexual relationships (1 item). The questionnaire has a 4-point scale. The total score is calculated as the sum of the subscale means and can range from 5 to 20. The minimal important difference ranges from 1.7 to 2.0 points.
Changes in snoring intensity measured with a Visual Analogue Scale (VAS) | 16 weeks of add-on therapy
  If patients have a bed partner, a standard 10-point VAS ranging from 0 (no snoring) to 10 (extreme snoring causing the bed partner to leave the bedroom or sleep separately) will be used to evaluate the subjective status of snoring during sleep. Heavy snoring corresponds to a snoring index of at least 7. A decrease of 3 points after treatment is considered significant. A satisfactory improvements is defined as a reduction to an index that is no longer experiences as bothersome (i.e. <3).
Incidence of adverse events | 16 weeks of add-on therapy
  Safety and tolerability of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Vanderveken, MD, PhD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium